CLINICAL TRIAL: NCT03331900
Title: A Phase 1 Single Ascending Dose Study of COR388 HCl
Brief Title: Study of COR388 HCl in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cortexyme Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: COR388-001
Record Dates: First submitted 2017-10-23; First posted 2017-11-06 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — COR388

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- COR388 TBD mg (Active Comparator)
  Interventions: Drug: COR388

INTERVENTIONS:
Drug: COR388 — Administered as oral capsule
  Arms: COR388 TBD mg
Drug: Placebo — Administered as oral capsule
  Arms: Placebo

SUMMARY:
The study is a randomized, double-blind, placebo-controlled, dose escalation, first-in-human trial of the safety and tolerability of COR388 HCl in healthy male and female subjects.

ELIGIBILITY:
Major Inclusion Criteria:

1. Males of reproductive potential must agree to use double-barrier contraceptive measures or avoid intercourse from Day -1 through 28 days after the dose of study drug;
2. Females of child-bearing potential must be non-lactating, have negative serum pregnancy test results at screening visit and Day 1; agree to use double-barrier contraceptive measures or avoid intercourse from Day -10 through 28 days after the dose of study drug;
3. Body mass index (BMI) ≥19 to ≤32 kg/m2;
4. Good health as determined by the absence of clinically significant deviation from normal, by medical history, physical examination, laboratory reports, and 12-lead electrocardiogram (ECG) prior to enrollment;
5. Non-smoker and non-tobacco user for a minimum of 3 months prior to screening and for the duration of the study;
6. Able to understand and willing to comply with all study requirements, and follow the study medication regimen.

Major Exclusion Criteria:

1. History or current evidence of cardiac, hepatic, renal, pulmonary, endocrine, neurologic, gastrointestinal, hematologic, oncologic, infectious, or psychiatric disease as determined by screening history, physical examination, laboratory reports, or 12-lead ECG;
2. Need for any concomitant medication (with the exception of hormonal contraceptives as allowed for females of child-bearing potential);
3. Use of any prescription drug within 14 days prior to the first dose of the study (with the exception of hormonal contraceptives for females of childbearing potential);
4. Use of any non-prescription drug and/or herbal supplements within 7 days prior to the first dose of the study;
5. History of significant allergic reaction to any drug;
6. Participation in another investigational new drug research study within the 30 days prior to the first dose of the study;
7. History of alcohol or drug abuse or dependence within 12 months of screening as determined by the Investigator;
8. Positive urine screen for prohibited drugs or positive alcohol screen on Day -1.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2018-02-20 (Actual); Study Completion 2018-04-02 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration curve (AUC) | 72 hours
  Analysis of AUC
Maximum observed plasma concentration (Cmax) | 72 hours
  Analysis of Cmax
Time of the first occurrence of the maximum observed plasma concentration (Tmax) | 72 hours
  Analysis of Tmax

SECONDARY OUTCOMES:
Incidence of treatment emergent adverse events | 72 Hours
  Assessment of the incidence and severity of treatment-emergent adverse events.
Changes in chemistry lab measures (Sodium [Na], Blood Urea Nitrogen [BUN], Calcium [Ca], Total bilirubin). | 72 hours
  Assessment of changes in serum chemistry measures.
Changes in hematology lab measures (RBC, Hgb, Hct). | 72 hours
  Assessment of changes in hematology measures.
Changes in urinalysis lab parameters (pH, specific gravity, glucose). | 72 hours
  Assessment of changes in urinalysis parameters.

CONTACTS AND LOCATIONS:
Locations (1):
- Medpace Clinical Pharmacology Unit, Cincinnati, Ohio, United States